CLINICAL TRIAL: NCT02532881
Title: Evaluation of a Video-based Internet Intervention as Preparation for Inpatient Psychosomatic Rehabilitation: A Randomized Controlled Trial
Brief Title: Evaluation of a Video-based Internet Intervention as Preparation for Inpatient Psychosomatic Rehabilitation
Acronym: Reh@:Info
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: University of Kaiserslautern-Landau (Other); Deutsche Rentenversicherung (Other)
Responsible Party: Principal Investigator, Dr. Rüdiger Zwerenz, Dr., Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RK-93184
Record Dates: First submitted 2015-07-30; First posted 2015-08-26 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Outcome Expectancy
MeSH Terms: interventions — Videotape Recording; Therapeutics

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as ususal (TAU) + Video Access (Experimental): Patients in this arm receive access to various videos on the study website as well as treatment as usual (written information provided by the clinic).
  Interventions: Other: Videos; Other: Treatment as usual
- Treatment as usual (TAU) (Placebo Comparator): Patients in this arm receive treatment as usual (written information provided by the clinic).
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Videos — Various videos showing four characteristic patient stories and five expert statements on special topics concerning inpatient psychosomatic rehabilitation.
  Arms: Treatment as ususal (TAU) + Video Access
Other: Treatment as usual — Treatment as usual

SUMMARY:
The purpose of this study is to determine the effect of an internet-based preparation on the outcome expectancy and treatment credibility of rehabilitants concerning inpatient psychosomatic rehabilitation. Both study groups receive the usual written information for preparation (TAU). The patients of the experimental group have access to various videos on the study website until their inpatient rehabilitation begins, the patients of the placebo group receive no special treatment. The investigators hypothesize that the experimental group gains more positive outcome expectancy and treatment credibility compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Authorized inpatient rehabilitation in one of the cooperation clinics
* Internet access

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Outcome expectancy measured with the "Credibility Expectancy Questionnaire" (CEQ) | Two weeks before inpatient rehabilitation (T1)

SECONDARY OUTCOMES:
Work-related therapy motivation measured with the "Work-Related Therapy Motivation Questionnaire" (FBTM) | Two weeks before inpatient rehabilitation (T1)
Treatment motivation measured with the "Questionnaire for Assessment of Rehabilitation Expectancy and Motivation" (FREM-17) and the "Patient Questionnaire for Assessment of Rehabilitation Motivation-20" (PAREMO-20) | Two weeks before inpatient rehabilitation (T1)
Functioning in everyday life measured with the "Indicators of Rehabilitation Status-24" (IRES-24) | At the end of inpatient rehabilitation, an expected average of six weeks after admission to inpatient rehabilitation (T2)
Satisfaction with inpatient rehabilitation measured with the "Patient Satisfaction Questionnaire-8" (ZUF-8) | At the end of inpatient rehabilitation, an expected average of six weeks after admission to inpatient rehabilitation (T2)
Depression and anxiety measured with the "Patient Health Questionnaire-4" (PHQ-4) | At the end of inpatient rehabilitation, an expected average of six weeks after admission to inpatient rehabilitation (T2)
Satisfaction with and usage of IP with a self devised questionnaire | Two weeks before inpatient rehabilitation (T1)
Perceived advantage of after care measured with a self devised questionnaire | Two weeks before inpatient rehabilitation (T1)
Internet usage and technology affinity measured with a self devised questionnaire | At study inclusion (T0)
Use of online clinic review portals and the cooperation clinics websites measured with a self devised questionnaire | Two weeks before inpatient rehabilitation (T1)
Treatments, especially rehabilitations, prior to this inpatient rehabilitation measured with a self devised questionnaire | At study inclusion (T0)
Subjective prognosis of work ability measured with the questionnaire "Subjective Prognosis of Work-Ability" (SPE) | At the end of inpatient rehabilitation, an expected average of six weeks after admission to inpatient rehabilitation (T2)
Treatment credibility measured with the "Credibility Expectancy Questionnaire" (CEQ) | Two weeks before inpatient rehabilitation (T1)
Mental condition "Indicators of Rehabilitation Status-24" (IRES-24) | At the end of inpatient rehabilitation, an expected average of six weeks after admission to inpatient rehabilitation (T2)

CONTACTS AND LOCATIONS:
Overall Officials: Rüdiger Zwerenz, Dr., Principal Investigator — University Medical Center, Department of Psychosomatic Medicine and Psychotherapy, Johannes Gutenberg University Mainz
Locations (5):
- Germany (5):
  - Center for Rehabilitation Bad Kissingen, Bad Kissingen, Bavaria
  - Psychosomatic Clinic Bad Neustadt, Bad Neustadt an der Saale, Bavaria
  - AHG Clinic for Psychosomatic Rehabilitation Bad Dürkheim, Bad Dürkheim, Rhineland-Palatinate
  - Knowledge Media Institute of the University of Koblenz-Landau, Koblenz, Rhineland-Palatinate
  - University Medical Center, Department of Psychosomatic Medicine and Psychotherapy, Johannes Gutenberg University, Mainz, Rhineland-Palatinate

REFERENCES:
- [Derived] Becker J, Beutel ME, Gerzymisch K, Schulz D, Siepmann M, Knickenberg RJ, Schmadeke S, Ferdinand P, Zwerenz R. Evaluation of a video-based Internet intervention as preparation for inpatient psychosomatic rehabilitation: study protocol for a randomized controlled trial. Trials. 2016 Jun 13;17(1):287. doi: 10.1186/s13063-016-1417-y. PMID 27296249